CLINICAL TRIAL: NCT01425190
Title: Assessment of the Pharmacokinetics of Boceprevir in Pediatric Subjects With Chronic Hepatitis C Genotype 1 (Phase 1b); Protocol No. P07614
Brief Title: Pharmacokinetics of Boceprevir in Pediatric Subjects With Chronic Hepatitis C Genotype 1 (P07614)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The US FDA and the EU CHMP provided guidance indicating preference for intereferon-free regimens in pediatric studies of HCV infection.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P07614; 2010-023498-20 (EudraCT Number); MK-3034-063 (Other: Merck)
Record Dates: First submitted 2011-08-26; First posted 2011-08-29 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1: Children 17 to ≥13 years (Experimental): Participants were administered a single dose of boceprevir powder mixed in a suitable vehicle such pudding or applesauce. The first 4 participants were treated with a 11.4 mg/kg dose of boceprevir powder. The dose/weight ratio may be adjusted for the next 12 participants based on the evaluation of the PK, safety, and tolerability data from the first 4 participants.
  Interventions: Drug: Boceprevir
- Cohort 2: Children <13 to ≥7 years (Experimental): Participants were administered a single dose of boceprevir powder mixed in a suitable vehicle such as pudding or applesauce. The first 4 participants were treated with boceprevir at a dose contingent on the PK and safety results in Cohort 1. The dose/weight ratio may be adjusted for the next 12 participants based on the evaluation of the PK, safety, and tolerability data from the first 4 participants.
  Interventions: Drug: Boceprevir
- Cohort 3: Children <7 to ≥3 years (Experimental): Participants were administered a single dose of boceprevir powder mixed in a suitable vehicle such as pudding or applesauce. The first 4 participants were treated with boceprevir at a dose contingent on the PK and safety results in Cohort 2. The dose/weight ratio may be adjusted for the next 12 participants based on the evaluation of the PK, safety, and tolerability data from the first 4 participants.
  Interventions: Drug: Boceprevir

INTERVENTIONS:
Drug: Boceprevir — Single dose of boceprevir powder prior to breakfast in a dosing vehicle of chocolate pudding (i.e., a mousse or custard), apple sauce, Nutella, fruit pudding such as strawberry, cherry, or raspberry pudding, or yogurt or a similar semi-solid product into which the boceprevir powder can be evenly stirred
  Other Names: SCH 503034

SUMMARY:
This is a study to determine the pharmacokinetics (PK) and weight-based dose of boceprevir following single oral dose administration in Chronic Hepatitis C Virus (HCV) pediatric participants.

ELIGIBILITY:
Inclusion Criteria:

* Documented chronic hepatitis C (CHC) genotype 1 infection
* Treatment naïve or failed previous interferon/ribavirin therapy (≥12 uninterrupted weeks)
* Weigh between 10 kg to 90 kg inclusive at screening and baseline (Day -1).
* Body Mass Index (BMI) from the 5th to the 95th percentile for the participant's age and gender, inclusive, per tables from the Center for Disease Control and Prevention, USA
* Use of acceptable methods of contraception for at least 3 months prior to baseline and continue on study

Exclusion Criteria:

* Co-infection with the human immunodeficiency virus (HIV) or hepatitis B virus (HBsAg positive).
* Treatment with ribavirin within 90 days, or any interferon-alfa within 30 days
* Discontinued from interferon treatment due to adverse events
* Currently receiving antiviral/immunomodulating therapy for hepatitis C
* Prior treatment with an HCV protease inhibitor
* Prior treatment with any known hepatotoxic agent (including herbal remedies)
* Use of investigational drugs within 30 days of enrollment into study
* Evidence of de-compensated liver disease including, but not limited to, a history or presence of clinical ascites, bleeding varices, or hepatic encephalopathy.
* Substance abuse (including but not limited to alcohol abuse, illicit drugs,

inhalational drugs, marijuana use, etc) any time prior to entry into the study

* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug.
* Pregnant or breastfeeding female
* Meeting any of the laboratory exclusion criteria

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2012-01-04 (Actual); Primary Completion 2013-03-20 (Actual); Study Completion 2013-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P07614&kw=P07614&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study originally intended to enroll 3 age-based pediatric cohorts. However the study was terminated after the completion of Cohort 1. No participants were enrolled in either Cohorts 2 or 3. Only data from Cohort 1 was collected.
Period: Overall Study
Arm/Group | Cohort 1: Children 17 to ≥13 Years | Cohort 2: Children <13 to ≥7 Years | Cohort 3: Children <7 to ≥3 Years
Started | 16 | 0 (The study was terminated prior to enrolling participants in Cohort 2.) | 0 (The study was terminated prior to enrolling participants in Cohort 3.)
Completed | 15 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Full dose not consumed. | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Population includes all participants in Cohort 1 that received boceprevir. The trial was terminated prior to enrolling participants in either Cohorts 2 or 3.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Children 17 to ≥13 Years | Cohort 2: Children <13 to ≥7 Years | Cohort 3: Children <7 to ≥3 Years | Total
Number analyzed (Participants) | 16 | 0 | 0 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 14.9 (1.2) |  |  | 14.9 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 |  |  | 7
  Male | 9 |  |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time Curve (AUC) From 0-Infinity of Single Dose Boceprevir
Description: Plasma concentrations of boceprevir were determined at 0 (pre-dose), 0.5, 1, 2, 2.5, 4.5, 5.5, 8, and 10 hours post dose.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 2.5, 4.5, 5.5, 8, and 10 hours post dose
Population: The Per Protocol (PP) population includes all participants who complied with the protocol sufficiently to ensure that data for this assessment were likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Mean (Full Range); unit: ng hr/mL
Arm/Group | Cohort 1: Children 17 to ≥13 Years | Cohort 2: Children <13 to ≥7 Years | Cohort 3: Children <7 to ≥3 Years
Number analyzed (Participants) | 14 | 0 | 0
ng hr/mL | 6660 [3860 to 10500] |  |

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Single Dose Boceprevir
Description: The maximum observed plasma concentration of boceprevir across sampling intervals was determined.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 2.5, 4.5, 5.5, 8, and 10 hours post dose
Population: as for outcome 1
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Cohort 1: Children 17 to ≥13 Years | Cohort 2: Children <13 to ≥7 Years | Cohort 3: Children <7 to ≥3 Years
Number analyzed (Participants) | 15 | 0 | 0
ng/mL | 1710 [985 to 2320] |  |

3. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of Single Dose Boceprevir
Description: The time at which the maximum plasma boceprevir concentration was observed.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 2.5, 4.5, 5.5, 8, and 10 hours post dose
Population: as for outcome 1
Measure: Mean (Full Range); unit: Hour
Arm/Group | Cohort 1: Children 17 to ≥13 Years | Cohort 2: Children <13 to ≥7 Years | Cohort 3: Children <7 to ≥3 Years
Number analyzed (Participants) | 15 | 0 | 0
Hour | 1.87 [0.4 to 4.5] |  |

4. Primary Outcome: Final Dose of Boceprevir By Age Group
Time Frame: Day 1
Population: This outcome measure could not be analyzed due to termination of the study prior to enrolling Cohorts 2 and 3.
Arm/Group | Cohort 1: Children 17 to ≥13 Years | Cohort 2: Children <13 to ≥7 Years | Cohort 3: Children <7 to ≥3 Years
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Nonserious adverse events (AEs) and serious AEs (SAEs) were collected during the time of boceprevir administration until the final PK sample was collected on Day 1.
Description: AEs were monitored in the All Subjects as Treated (all boceprevir-treated participants) population.
Arm/Group | Cohort 1: Children 17 to ≥13 Years | Cohort 2: Children <13 to ≥7 Years | Cohort 3: Children <7 to ≥3 Years
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 6/16 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Children 17 to ≥13 Years (N=16) | Cohort 2: Children <13 to ≥7 Years (N=0) | Cohort 3: Children <7 to ≥3 Years (N=0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Children 17 to ≥13 Years (N=16) | Cohort 2: Children <13 to ≥7 Years (N=0) | Cohort 3: Children <7 to ≥3 Years (N=0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication.